CLINICAL TRIAL: NCT04938440
Title: Assessment of the Effectiveness of Updated Educational Materials on Prescribers' Knowledge and Behavior With Respect to Risks Associated With INSTANYL® Off-Label Use
Brief Title: Assessment of Updated Educational Materials for Instanyl®
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Instanyl-5002
Record Dates: First submitted 2021-06-23; First posted 2021-06-24 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Pain; Cancer Pain
Keywords: Drug Therapy
MeSH Terms: conditions — Pain; Cancer Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prescribers of Instanyl®: Healthcare professionals (Oncologists, oncoradiologists, anaesthesiologists, pain management prescribers, palliative care prescribers, internal medicine prescribers, general practitioners and other specialties) who are current and potential prescribers of Instanyl® will be assessed before and after the distribution of the updated EMs via web-based survey questionnaire.

SUMMARY:
The purpose of the Instanyl study is to learn how much doctors know and understand about Instanyl® before and after they receive updated educational information, including the risks of its unapproved use. In this study, the doctors will complete two surveys: one three months before they receive the updated educational information, and one about six months after they receive this information. They will answer questions about their prescribing behavior plus their knowledge of Instanyl® including any risks.

DETAILED DESCRIPTION:
This is a non-interventional, observational, cross-sectional study of prescribers of Instanyl®.

This study will assess the prescribers' awareness of the updated EMs and changes in prescribers' knowledge and understanding of the key information contained in the updated EMs. The study will enroll approximately 259 prescribers. The first survey (pre-EM survey) will be conducted three months before the distribution of updated EMs, second survey (post-EM survey) will be conducted six months following the distribution of updated EMs.

The data will be collected, through a self-administered web-based questionnaire. All participants will be enrolled in a single observational group:

• Prescriber of Instanyl®

This multi-center study will be conducted in France, the Netherlands, and Poland. The overall duration of the study will be approximately 22 months.

ELIGIBILITY:
Inclusion Criteria:

1. Specialists of any of those medical specialties targeted for the EMs as agreed with each national competent authority. The foreseen specialties include the following (subject to changes after the EM distribution plan is completed and agreed with national competent authorities):

   * Oncologists and oncoradiologists
   * Anaesthesiologists
   * Pain management prescribers
   * Palliative care prescribers
   * Internal medicine prescribers
   * General practitioner (GPs)
   * Other specialties may be locally included such as hematology. Current and potential prescribers may vary between country; thus, some countries may have modified lists of target specialties.
2. Physicians who have prescribed Instanyl® in the past 12 months (pre-EM survey) or since the updated EMs (post-EM survey) and who intend to prescribe Instanyl® in the following months after each survey.

Exclusion Criteria:

1. Physicians who may have a conflict of interest (that is, prescribers employed by regulatory bodies, pharmaceutical industries).
2. Inactive or retired prescribers.
3. Physicians who did not prescribe Instanyl® in the past 12 months (pre-EM survey) or since the updated EMs are distributed (post-EM survey) and do not foresee treating a participants with Instanyl® in the following 12 months, regardless of whether they have prescribed Instanyl® before.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prescribers of Instanyl® will be assessed before and after the distribution of the updated EMs.
Sampling Method: Non-Probability Sample
Enrollment: 536 (Actual)
Dates: Start 2022-02-18 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2023-02-06 (Actual)

PRIMARY OUTCOMES:
Percentage of Prescribers With Awareness of Updated Educational Materials (EMs) Based on Post-EM Questionnaire Survey | Up to 6 months (Post-EM Survey)
Percentage of Prescribers With Change in Knowledge and Understanding of Key Safety Information Contained in Updated EMs Based on Pre-EM to Post-EM Questionnaire Survey | Up to 9 months (Pre-EM to Post-EM survey)
Percentage of Prescribers With Change in Self-Reported Behavior Prescribing Based on Pre-EM to Post-EM Questionnaire Survey | Up to 9 months (Pre-EM to Post-EM survey)
Number of Reasons for Off-label Prescription | Up to 3 months (Pre-EM survey)
Number of Prescribers With Awareness of the Profile of Patients at Risk of Misuse and Addiction | Up to 6 months (Post-EM Survey)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Central Contact, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/60d5b75bef0b71001e743df7